CLINICAL TRIAL: NCT06413537
Title: A Phase 2a, Randomized, Double-Blinded, Study Evaluating the Neurophysiologic vs Clinical Effects of Single-Dose SPG601 and Placebo in Adult Men With Fragile X Syndrome
Brief Title: Study of SPG601 in Adult Men With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spinogenix (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPG601-01
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; Fragile X Chromosome; cognitive outcomes
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Active SPG601 to be administered to participants with Fragile X Syndrome (Active Comparator): Participants with Fragile X Syndrome will be randomized to receive SPG601 or placebo (8 capsules of 100 mg) one time on days 1 and 8 of the study.
  Interventions: Drug: SPG601
- Placebo Comparator: Placebo comparator to be administered to participants with Fragile X Syndrome (Placebo Comparator): Participants with Fragile X Syndrome will be randomized to receive SPG601 or placebo (8 capsules of 100 mg) one time on days 1 and 8 of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPG601 — synthetic small molecule
  Arms: Experimental: Active SPG601 to be administered to participants with Fragile X Syndrome
Drug: Placebo — Placebo
  Arms: Placebo Comparator: Placebo comparator to be administered to participants with Fragile X Syndrome

SUMMARY:
This Phase 2 study described herein will evaluate the safety, efficacy, tolerability, pharmacokinetics and pharmacodynamics of SPG601 in adult men with Fragile X syndrome.

DETAILED DESCRIPTION:
This study is a Phase 2 randomized, double blind, placebo-controlled, cross over, single dose of SPG601 and matching Placebo in patients with Fragile X syndrome.

This study will entail 2 in person clinic visits to administer oral doses of SPG601 or matching placebo. Participants will receive a dose of either SPG601 or placebo at first visit, and will cross over to receive the other product at the second visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 18 to 45 years
* Diagnosis of Fragile X as confirmed with genetic testing
* Patient must have caregiver
* Must be in good health with no significant medical history
* Clinical laboratory values within normal range or < 1.2 times ULN
* Contraceptive use by men or women consistent with local regulations
* Able and willing to provide written informed consent
* Stable dosing of psychotropic drugs for at least 4 weeks

Exclusion Criteria:

* Any physical or psychological condition that prohibits study completion
* Uncontrolled seizures or history of epilepsy with a seizure in the past 6 months.
* Auditory or visual impairments that can not be corrected
* History of suicidal behavior or suicidal ideation
* Screening vital signs that are abnormal per protocol specification
* ECG that are clinically significant abnormal
* History of substance abuse or dependence within 6 months
* Other investigational products within 30 days

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions Improvement scale as determined by the treating clinician | 15 days
  Change in clinician rated measures on scale of 1 to 7, higher value indicates more severe symptom presentation
Clinical Global Impressions Improvement scale as determined by the caregiver | 15 days
  Change in caregiver rated measures on scale of 1 to 7, higher value indicates more severe symptom presentation
Visual Analog scale as determined by the patient caregiver | 15 days
  Change in notation on Visual Analog scale as determined by the patient caregiver. Rater will indicate on linear measurement scale of 1 to 100 centimeters, with higher score indicating more severe symptoms
Change in auditory response to chirp stimulus | 15 days
  Auditory test will be evaluated for difference in responses to stimuli.

SECONDARY OUTCOMES:
Change in attention and inhibition symptoms | 15 days
  KiTAP Tests of Attentional Performance for Children, to measure alertness and assessments of visual reactions
Change in cognitive outcomes measured by NIH Cognitive Toolbox | 15 days
  National Institute of Health (NIH)- Toolbox Cognitive Battery (TCB):
  A series of tests will be conducted to assess reading, vocabulary, and speed matching. These tests are scored from zero to 100. A higher score indicate better performance.
Change in eye tracking for social gaze | 15 days
  This test will measure eye tracking and movement in response to stimuli, and social gaze version, with a Likert scale of 1-5 for behavior rating.
Change in memory and cognitive assessment with RBANS list learning. | 15 days
  RBANS (Repeatable Battery for the Assessment of Neuropsychological Status) is scored from -4 to 4, with higher values indicate higher memory and cognitive assessment
Change in auditory response to steady state auditory stimuli | 15 days
  Auditory test will be evaluated for difference in responses to stimuli.
Change in eye tracking measured by electroretinography | 15 days
  This test will measure the electrical activity in the retina in response to stimuli
Safety and tolerability of SPG601 in patients with Fragile X Syndrome | 15 days
  Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Erickson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States